CLINICAL TRIAL: NCT01201954
Title: Pain Relief of Newborn Preterm Infants During Endotracheal Suctioning: a Randomized Clinical Trial
Brief Title: Pain Relief of Newborn Preterm Infants During Endotracheal Suctioning
Acronym: PRPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Rita de Cássia de Albuquerque Almeida, Pós-graduação em Saúde da Criança e do Adolescente - UFPE
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SACAROSE01
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2010-09

CONDITIONS: Pain
Keywords: pain; sucrose; newborn; mechanical ventilation
MeSH Terms: conditions — Pain | interventions — Sucrose; Sugars

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sucrose (Active Comparator): 0,5 ml/kg of sucrose administered 2 minutes prior the procedure
  Interventions: Drug: sucrose
- sterile water (Placebo Comparator): 0,5 ml/kg of sterile water administered 2 minutes prior the procedure
  Interventions: Drug: sucrose

INTERVENTIONS:
Drug: sucrose — oral sucrose solution, 24%, 0,5 ml/kg, 2 minutes before start the suctioning sterile water, 0,5 ml/kg, 2 minutes before start the suctioning
  Other Names: sugar

SUMMARY:
Evaluate the effectiveness of the use of a 24% sucrose solution for pain management of preterm infants during endotracheal suctioning.

DETAILED DESCRIPTION:
Many infants admitted to neonatal intensive care unit (NICU) undergo repeated invasive procedures. Recent studies have shown that the oral sucrose administration to neonates is safe and effective for pain relief during heel stick and venipuncture.Most data suggest the investigation of the effect of sucrose in other painful procedures such as in ventilated newborns.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants
* over 12 hours of life
* intubated
* clinically stable
* without use of analgesics or sedatives

Exclusion Criteria:

* preterms with congenital malformations
* preterms with genetic syndromes
* preterms with Apgar score at 5´<7
* preterms with meningitis
* preterms with diagnosed of necrotizing enterocolitis Ouvir Ler foneticamente

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
clinical pain score | within the first twelve hours after clinical stabilization, the PIPP will be done.
  The tool that will be used is PIPP = Premature Infant Pain Profile. This avaliation begins prior to suctioning until 30 seconds after suctioning. Each infant will be avaliated 2 times (with sucrose and with placebo). The 2 avaliations in the same day.

CONTACTS AND LOCATIONS:
Overall Officials: Rita A Almeida, postgraduate, Principal Investigator — Universidade Federal de Pernambuco; Sônia B Coutinho, Dr., Study Director — Universidade Federal de Pernambuco; Pedro I Lira, Dr., Study Director — Universidade Federal de Pernambuco
Locations (1):
- Hospital Agamenon Magalhães, Hospital Barão de Lucena, Recife, Pernambuco, Brazil